CLINICAL TRIAL: NCT02293902
Title: A Randomized, Double-blind, Multicenter Study With a Placebo-controlled Period Assessing the Efficacy and Safety of Sarilumab Added to Methotrexate (MTX) in Japanese Patients With Moderately to Severely Active Rheumatoid Arthritis Who Are Inadequate Responders to MTX Therapy
Brief Title: A Study Assessing the Efficacy and Safety of Sarilumab Added to MTX in Japanese Patients With Moderately to Severely Active Rheumatoid Arthritis (SARIL-RA-KAKEHASI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC14059; U1111-1155-7401 (Other: UTN)
Record Dates: First submitted 2014-11-13; First posted 2014-11-19 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab; Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: Yes

ARMS (4):
- Sarilumab 150 mg/150 mg (Experimental): Sarilumab 150 mg subcutaneous (SC) injection once every 2 weeks (q2w) in combination with MTX and folic acid in double-blind period up to Week 24 followed by single-blind period in which participants continued with the same treatment up to Week 52. Participants with inadequate response (defined as less than 20% improvement from baseline on 2 consecutive visits [at least 4 weeks apart] in either tender joint count [TJC] or swollen joint count [SJC], or with any other clear lack of efficacy based on investigator's judgment) by Week 16, were rescued with open label sarilumab 200 mg q2w treatment.
  Interventions: Drug: Sarilumab SAR153191 (REGN88); Drug: Methotrexate; Drug: Folic acid
- Sarilumab 200 mg/200 mg (Experimental): Sarilumab 200 mg SC injection q2w in combination with MTX and folic acid in double-blind period up to Week 24 followed by single-blind period in which participants continued with the same treatment up to Week 52. Participants with inadequate response (defined as less than 20% improvement from baseline on 2 consecutive visits [at least 4 weeks apart] in either TJC or SJC, or with any other clear lack of efficacy based on investigator's judgment) by Week 16, were rescued with open label sarilumab 200 mg q2w treatment.
  Interventions: Drug: Sarilumab SAR153191 (REGN88); Drug: Methotrexate; Drug: Folic acid
- Placebo/Sarilumab 150 mg (Placebo Comparator): Placebo (for sarilumab) SC injection q2w in combination with MTX and folic acid in double-blind period up to Week 24 followed by a single-blind period in which participants were switched and received sarilumab 150 mg SC injection q2w in combination with MTX and folic acid up to Week 52. Participants with inadequate response (defined as less than 20% improvement from baseline on 2 consecutive visits [at least 4 weeks apart] in either TJC or SJC, or with any other clear lack of efficacy based on Investigator's judgment) by Week 16, were rescued with open label sarilumab 200 mg q2w treatment.
  Interventions: Drug: Sarilumab SAR153191 (REGN88); Other: Placebo (for sarilumab); Drug: Methotrexate; Drug: Folic acid
- Placebo/Sarilumab 200 mg (Placebo Comparator): Placebo (for sarilumab) SC injection q2w in combination with MTX and folic acid in double-blind period up to Week 24 followed by a single-blind period in which participants were switched and received sarilumab 200 mg SC injection q2w in combination with MTX and folic acid up to Week 52. Participants with inadequate response (defined as less than 20% improvement from baseline on 2 consecutive visits [at least 4 weeks apart] in either TJC or SJC, or with any other clear lack of efficacy based on Investigator's judgment) by Week 16, were rescued with open label sarilumab 200 mg q2w treatment.
  Interventions: Drug: Sarilumab SAR153191 (REGN88); Other: Placebo (for sarilumab); Drug: Methotrexate; Drug: Folic acid

INTERVENTIONS:
Drug: Sarilumab SAR153191 (REGN88) — Pharmaceutical form: solution for injection Route of administration: subcutaneous
Other: Placebo (for sarilumab) — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Arms: Placebo/Sarilumab 150 mg; Placebo/Sarilumab 200 mg
Drug: Methotrexate — Dispensed according to local practice.
Drug: Folic acid — Dispensed according to local practice.

SUMMARY:
Primary Objective:

-To demonstrate that sarilumab added to methotrexate (MTX) reduce signs and symptoms of rheumatoid arthritis (RA) in Japanese RA participants with an inadequate response to MTX.

Secondary Objective:

-To assess the safety of sarilumab added to MTX in Japanese RA participants with an inadequate response to MTX.

DETAILED DESCRIPTION:
The total duration of study was expected up to 62 weeks (screening period of 4 weeks, treatment period of 52 weeks, and a 6-week post treatment observation).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of RA, according to the American College of Rheumatology/The European League Against Rheumatism (ACR/EULAR) 2010 Rheumatoid Arthritis Classification Criteria with >=3 months disease duration.
* Moderately to severely active RA defined as:
* At least 8 of 68 tender joints and 6 of 66 swollen joints at screening visit.
* High sensitivity C-Reactive Protein (hs-CRP) >=6mg/L at screening visit.

Exclusion criteria:

* Participants <20 or >75 years of age.
* Treatment with any Disease-modifying antirheumatic drug (DMARD) other than MTX or biologic agent without the appropriate off-drug period prior to screening.
* Prior treatment with anti-interleukin-6 (anti-IL-6) or anti-interleukin-6 receptor (IL-6R) antagonist therapies, including but not limited to tocilizumab or sarilumab.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (96):
- Japan (96):
  - Investigational Site Number 392010, Asahi-Shi
  - Investigational Site Number 392001, Asahikawa-Shi
  - Investigational Site Number 392035, Asahikawa-Shi
  - Investigational Site Number 392070, Beppu-Shi
  - Investigational Site Number 392036, Chiba
  - Investigational Site Number 392083, Chūōku
  - Investigational Site Number 392047, Fuchu-Shi
  - Investigational Site Number 392004, Fukui-shi
  - Investigational Site Number 392007, Fukuoka
  - Investigational Site Number 392038, Fukuoka
  - Investigational Site Number 392039, Fukuoka
  - Investigational Site Number 392078, Fukushima
  - Investigational Site Number 392054, Funabashi-Shi
  - Investigational Site Number 392015, Hachioji-Shi
  - Investigational Site Number 392085, Hannan-Shi
  - Investigational Site Number 392091, Hiroshima
  - Investigational Site Number 392098, Hiroshima
  - Investigational Site Number 392009, Hitachi-Naka
  - Investigational Site Number 392011, Hitachi-Naka
  - Investigational Site Number 392030, Ichinomiya-Shi
  - Investigational Site Number 392002, Iizuka-Shi
  - Investigational Site Number 392019, Kagoshima
  - Investigational Site Number 392066, Kamakura-Shi
  - Investigational Site Number 392086, Kamogawa-Shi
  - Investigational Site Number 392050, Kato-Shi
  - Investigational Site Number 392037, Kawachi-Nagano-Shi
  - Investigational Site Number 392093, Kawagoe-Shi
  - Investigational Site Number 392099, Kawasaki-Shi
  - Investigational Site Number 392016, Kirishima-Shi
  - Investigational Site Number 392013, Kitakyushu-Shi
  - Investigational Site Number 392024, Kitakyushu-Shi
  - Investigational Site Number 392045, Kitakyushu-Shi
  - Investigational Site Number 392063, Kiyose-Shi
  - Investigational Site Number 392051, Kobe
  - Investigational Site Number 392097, Kochi
  - Investigational Site Number 392040, Koushi-Shi
  - Investigational Site Number 392069, Kumamoto
  - Investigational Site Number 392089, Kurashiki-Shi
  - Investigational Site Number 392065, Kushiro
  - Investigational Site Number 392026, Matsuyama
  - Investigational Site Number 392081, Matsuyama
  - Investigational Site Number 392094, Matsuyama
  - Investigational Site Number 392042, Meguro-Ku
  - Investigational Site Number 392082, Meguro-Ku
  - Investigational Site Number 392012, Mito
  - Investigational Site Number 392034, Miyagi-Gun
  - Investigational Site Number 392053, Morioka
  - Investigational Site Number 392032, Nagano
  - Investigational Site Number 392064, Nagasaki
  - Investigational Site Number 392043, Nagoya
  - Investigational Site Number 392056, Nagoya
  - Investigational Site Number 392076, Nagoya
  - Investigational Site Number 392080, Nagoya
  - Investigational Site Number 392031, Nakano
  - Investigational Site Number 392046, Narashino-Shi
  - Investigational Site Number 392067, Narashino-Shi
  - Investigational Site Number 392044, Nishinomiya-Shi
  - Investigational Site Number 392062, Okayama
  - Investigational Site Number 392008, Omura-Shi
  - Investigational Site Number 392057, Osaka
  - Investigational Site Number 392060, Osaka
  - Investigational Site Number 392061, Osaka
  - Investigational Site Number 392096, Osaka
  - Investigational Site Number 392027, Osaki-Shi
  - Investigational Site Number 392059, Ōita
  - Investigational Site Number 392049, Sagamihara-Shi
  - Investigational Site Number 392072, Saitama-Shi
  - Investigational Site Number 392075, Sakaishi
  - Investigational Site Number 392014, Sapporo
  - Investigational Site Number 392068, Sapporo
  - Investigational Site Number 392073, Sapporo
  - Investigational Site Number 392006, Sasebo-Shi
  - Investigational Site Number 392021, Sendai
  - Investigational Site Number 392022, Sendai
  - Investigational Site Number 392033, Sendai
  - Investigational Site Number 392071, Sendai
  - Investigational Site Number 392100, Sendai
  - Investigational Site Number 392029, Shizuoka
  - Investigational Site Number 392025, Sumida-Ku
  - Investigational Site Number 392092, Sumida-Ku
  - Investigational Site Number 392023, Takaoka-Shi
  - Investigational Site Number 392095, Takarazuka-Shi
  - Investigational Site Number 392020, Takasaki-Shi
  - Investigational Site Number 392088, Takatsuki-Shi
  - Investigational Site Number 392018, Tokorozawa-Shi
  - Investigational Site Number 392003, Tomakomai-Shi
  - Investigational Site Number 392005, Tomakomai-Shi
  - Investigational Site Number 392077, Tonami-Shi
  - Investigational Site Number 392052, Toshima-Ku
  - Investigational Site Number 392058, Toyama
  - Investigational Site Number 392055, Toyonaka-Shi
  - Investigational Site Number 392074, Urasoe-Shi
  - Investigational Site Number 392079, Urayasu-Shi
  - Investigational Site Number 392048, Yokohama
  - Investigational Site Number 392090, Yokohama
  - Investigational Site Number 392101, Yokohama

REFERENCES:
- [Derived] Tanaka Y, Takahashi T, Van Hoogstraten H, Praestgaard A, Kato N, Kameda H. Haemoglobin changes and disease activity in Japanese patients with rheumatoid arthritis treated with sarilumab. Clin Exp Rheumatol. 2023 May;41(5):1129-1139. doi: 10.55563/clinexprheumatol/jq9u8f. Epub 2022 Oct 28. PMID 36305354
- [Derived] Tanaka Y, Wada K, Takahashi Y, Hagino O, van Hoogstraten H, Graham NMH, Kameda H. Sarilumab plus methotrexate in patients with active rheumatoid arthritis and inadequate response to methotrexate: results of a randomized, placebo-controlled phase III trial in Japan. Arthritis Res Ther. 2019 Mar 20;21(1):79. doi: 10.1186/s13075-019-1856-4. PMID 30894208

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 95 centers in Japan between 06 November 2014 and 28 October 2016. A total of 388 participants were screened, of whom 243 participants were randomized and 145 were screen failures.
Pre-assignment Details: Participants were randomized to receive sarilumab 150 mg, 200 mg or placebo in a double-blind period up to Week 24 followed by single-blind period during which participants originally given placebo were switched to sarilumab 150 mg or 200 mg; those originally given 150 mg, 200 mg in double-blind period, continued with same treatment up to Week 52.
Groups:
- Placebo: Placebo (for sarilumab) subcutaneous (SC) injection once every 2 weeks (q2w) in combination with methotrexate (MTX) and folic acid in double-blind period up to Week 24. Participants with inadequate response by Week 16 were rescued with open label sarilumab 200 mg q2w treatment.
- Sarilumab 150 mg/150 mg: Sarilumab 150 mg SC injection q2w in combination with MTX and folic acid in double-blind period up to Week 24 followed by single-blind period in which participants continued with the same treatment up to Week 52. Participants with inadequate response by Week 16 were rescued with open label sarilumab 200 mg q2w treatment.
- Sarilumab 200 mg/200 mg: Sarilumab 200 mg SC injection q2w in combination with MTX and folic acid in double-blind period up to Week 24 followed by single-blind period in which participants continued with the same treatment up to Week 52. Participants with inadequate response by Week 16 were rescued with open label sarilumab 200 mg q2w treatment.
- Placebo/Sarilumab 150 mg: Participants who completed placebo (for sarilumab) treatment up to Week 24, were switched and received sarilumab 150 mg SC injection q2w in combination with MTX and folic acid in single-blind period up to Week 52. Participants with inadequate response by Week 16 were rescued with open label sarilumab 200 mg q2w treatment.
- Placebo/Sarilumab 200 mg: Participants who completed placebo (for sarilumab) treatment up to Week 24, were switched and received sarilumab 200 mg SC injection q2w in combination with MTX and folic acid in single-blind period up to Week 52. Participants with inadequate response by Week 16 were rescued with open label sarilumab 200 mg q2w treatment.
Period: Double-Blind Period (Up to Week 24)
Arm/Group | Placebo | Sarilumab 150 mg/150 mg | Sarilumab 200 mg/200 mg | Placebo/Sarilumab 150 mg | Placebo/Sarilumab 200 mg
Started | 82 | 81 | 80 | 0 | 0
Treated | 81 | 81 | 80 | 0 | 0
Rescued (Included both participants who completed and did not complete the study.) | 44 | 6 | 8 | 0 | 0
Completed | 71 (42 rescued and 29 not rescued completed.) | 74 (6 rescued and 68 not rescued completed.) | 70 (8 rescued and 62 not rescued completed.) | 0 | 0
Not Completed | 11 | 7 | 10 | 0 | 0
Not completed — Adverse Event | 5 | 6 | 8 | 0 | 0
Not completed — Lack of Efficacy | 5 | 1 | 2 | 0 | 0
Not completed — Randomized but not Treated | 1 | 0 | 0 | 0 | 0
Period: Single-Blind Period (Week 25 to Week 52)
Arm/Group | Placebo | Sarilumab 150 mg/150 mg | Sarilumab 200 mg/200 mg | Placebo/Sarilumab 150 mg | Placebo/Sarilumab 200 mg
Started | 0 | 74 (68 participants not rescued continued same treatment and 6 rescued continued open label treatment.) | 70 (62 participants not rescued continued same treatment and 8 rescued continued open label treatment.) | 34 (14 participants not rescued were switched and 20 rescued continued open label treatment.) | 37 (15 participants not rescued were switched and 22 rescued continued open label treatment.)
Completed | 0 | 66 (5 rescued and 61 not rescued completed.) | 68 (8 rescued and 60 not rescued completed.) | 33 (20 rescued and 13 not rescued completed.) | 31 (18 rescued and 13 not rescued completed.)
Not Completed | 0 | 8 | 2 | 1 | 6
Not completed — Adverse Event | 0 | 7 | 1 | 1 | 6
Not completed — Lack of Efficacy | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population which included all participants who had been allocated to a randomized treatment regardless of whether the treatment was actually administered.
Groups:
- Placebo: Placebo (for sarilumab) SC injection once q2w in combination with MTX and folic acid in double-blind period up to Week 24. Participants with inadequate response by Week 16 were rescued with open label sarilumab 200 mg q2w treatment.
- Sarilumab 150 mg/150 mg: Sarilumab 150 mg SC injection q2w in combination with MTX and folic acid in double-blind period up to Week 24 followed by single-blind period in which participants continued with the same treatment up to Week 52. Participants with inadequate response by Week 16 were rescued with open label sarilumab 200 mg q2w treatment .
- Sarilumab 200 mg/200 mg: Sarilumab 200 mg SC injection q2w in combination with MTX and folic acid in double-blind period up to Week 24 followed by single-blind period in which participants continued with the same treatment up to Week 52. Participants with inadequate response by Week 16 were rescued with open label sarilumab 200 mg q2w treatment .
- Total: Total of all reporting groups
Arm/Group | Placebo | Sarilumab 150 mg/150 mg | Sarilumab 200 mg/200 mg | Total
Number analyzed (Participants) | 82 | 81 | 80 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (11.5) | 56.1 (9.5) | 55.3 (11.0) | 54.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 63 | 61 | 189
  Male | 17 | 18 | 19 | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20 (ACR20) Response at Week 24
Description: American College of Rheumatology (ACR) response is a composite rating scale that includes 7 variables: tender joints count (TJC [68 joints]); Swollen joints count (SJC [66 joints]); levels of an acute phase reactant (high sensitivity C-reactive protein [hs-CRP level]); participant's assessment of pain (measured on 0 [no pain]-100 mm [worst pain] visual analog scale [VAS]); participant's global assessment of disease activity (measured on 0 [no arthritis activity]-100 mm [maximal arthritis activity] VAS); physician's global assessment of disease activity (measured on 0 [no arthritis activity]-100 mm [maximal arthritis activity] VAS); participant's assessment of physical function (measured by health assessment questionnaire disability index [HAQ-DI], with scoring range of 0 [better health] - 3 [worst health]). ACR20 response was defined as achieving at least 20% improvement in both TJC and SJC, and at least 20% improvement in at least 3 of the 5 other assessments.
Time Frame: Week 24
Population: Analysis was performed on modified intent-to-treat (mITT) population which included all randomized participants who received at least one dose of investigational medicinal product (IMP) and had an evaluable primary endpoint, irrespective of compliance with the study protocol and procedures.
Measure: Number; unit: percentage of participants
Groups:
- Sarilumab 150 mg: Sarilumab 150 mg SC injection q2w in combination with MTX and folic acid in double-blind period up to Week 24. Participants with inadequate response by Week 16 were rescued with open label sarilumab 200 mg q2w treatment.
- Sarilumab 200 mg: Sarilumab 200 mg SC injection q2w in combination with MTX and folic acid in double-blind period up to Week 24. Participants with inadequate response by Week 16 were rescued with open label sarilumab 200 mg q2w treatment.
Arm/Group | Placebo | Sarilumab 150 mg | Sarilumab 200 mg
Number analyzed (Participants) | 81 | 81 | 80
percentage of participants | 14.8 | 67.9 | 57.5
Statistical Analysis 1: Comparison: Placebo vs Sarilumab 150 mg; Analysis was performed using Cochran-Mantel-Haenszel (CMH) test stratified by prior biologic use (Yes, No) and weight at screening (<55 kg, >=55 kg); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Odds Ratio (OR) = 12.185, 95% CI 2-sided [5.583 to 26.594]; Placebo vs. Sarilumab 150 mg
Statistical Analysis 2: Comparison: Placebo vs Sarilumab 200 mg; Analysis was performed using CMH test stratified by prior biologic use (Yes, No) and weight at screening (<55 kg, >=55 kg); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Odds Ratio (OR) = 7.227, 95% CI 2-sided [3.446 to 15.158]; Placebo vs. Sarilumab 200 mg

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after informed consent form is signed. AE includes serious as well as non-serious AEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, In-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. Any AEs that developed or worsened or became serious during double-blind on-treatment period, single-blind on-treatment period up to 6-week post-treatment follow-up period (up to Week 58) were considered treatment-emergent.
Time Frame: For placebo arm: Baseline up to Week 24; For sarilumab 150 mg/150 mg, sarilumab 200 mg/200 mg and sarilumab rescue arm: Baseline up to Week 58; For placebo/sarilumab 150 mg and placebo/sarilumab 200 mg arm: Week 25 up to Week 58
Population: Analysis was performed on safety population which included all randomized participants who actually received at least one dose or a partial dose of IMP.
Measure: Number; unit: participants
Groups:
- Placebo: Placebo (for sarilumab) SC injection once q2w in combination with MTX and folic acid in double-blind period up to Week 24.
- Sarilumab 150 mg/150 mg: Sarilumab 150 mg SC injection q2w in combination with MTX and folic acid in double-blind period up to Week 24 followed by single-blind period in which participants continued with the same treatment up to Week 52.
- Sarilumab 200 mg/200 mg: Sarilumab 200 mg SC injection q2w in combination with MTX and folic acid in double-blind period up to Week 24 followed by single-blind period in which participants continued with the same treatment up to Week 52.
- Placebo/Sarilumab 150 mg: Participants who completed placebo (for sarilumab) treatment up to Week 24, were switched and received sarilumab 150 mg SC injection q2w in combination with MTX and folic acid in single-blind period up to Week 52.
- Placebo/Sarilumab 200 mg: Participants who completed placebo (for sarilumab) treatment up to Week 24, were switched and received sarilumab 200 mg SC injection q2w in combination with MTX and folic acid in single-blind period up to Week 52.
- Sarilumab Rescue: Participants who received either placebo or sarilumab 150 mg or 200 mg and had inadequate response (defined as less than 20% improvement from baseline on 2 consecutive visits [at least 4 weeks apart] in either TJC or SJC, or with any other clear lack of efficacy based on Investigator's judgment) by Week 16, were rescued with open label sarilumab 200 mg q2w treatment up to Week 52.
Arm/Group | Placebo | Sarilumab 150 mg/150 mg | Sarilumab 200 mg/200 mg | Placebo/Sarilumab 150 mg | Placebo/Sarilumab 200 mg | Sarilumab Rescue
Number analyzed (Participants) | 81 | 81 | 80 | 14 | 15 | 58
participants
  Treatment Emergent AEs | 49 | 76 | 71 | 12 | 13 | 54
  Treatment Emergent SAEs | 6 | 8 | 5 | 0 | 2 | 4

3. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Abnormalities
Description: Criteria for potentially clinically significant vital sign abnormalities:
  * Systolic blood pressure supine (SBP[S]): <=95 mmHg and decrease from baseline (DFB) >=20 mmHg; >=160 mmHg and increase from baseline (IFB) >=20 mmHg
  * Diastolic blood pressure supine (DBP[S]): <=45 mmHg and DFB >=10 mmHg; >=110 mmHg and IFB >=10 mmHg
  * Orthostatic systolic blood pressure (SBP[O]): <=-20 mmHg
  * Orthostatic diastolic blood pressure (DBP[O]): <=-10 mmHg
  * Heart rate supine (HR[S]): <=50 beats per minute (bpm) and DFB >=20 bpm; >=120 bpm and IFB >=20 bpm
  * Weight: >=5% DFB; >=5% IFB
Time Frame: as for outcome 2
Population: Analysis was performed on safety population.
Measure: Number; unit: participants
Arm/Group | Placebo | Sarilumab 150 mg/150 mg | Sarilumab 200 mg/200 mg | Placebo/Sarilumab 150 mg | Placebo/Sarilumab 200 mg | Sarilumab Rescue
Number analyzed (Participants) | 81 | 81 | 80 | 14 | 15 | 58
participants
  SBP(S) <=95 mmHg and DFB >=20 mmHg | 2 | 4 | 1 | 0 | 0 | 0
  SBP(S) >=160 mmHg and IFB >=20 mmHg | 2 | 5 | 5 | 0 | 1 | 8
  DBP(S) <=45 mmHg and DFB >=10 mmHg | 1 | 1 | 1 | 0 | 0 | 0
  DBP(S)>=110 mmHg and IFB >=10 mmHg | 0 | 1 | 0 | 0 | 0 | 0
  SBP(O) <=-20 mmHg | 8 | 21 | 23 | 2 | 2 | 12
  DBP(O) <=-10 mmHg | 8 | 17 | 12 | 0 | 1 | 10
  HR(S) <=50 bpm and DFB >=20 bpm | 0 | 4 | 1 | 0 | 0 | 1
  HR(S) >=120 bpm and IFB >=20 bpm | 1 | 0 | 0 | 0 | 0 | 0
  Weight >=5% DFB: number analyzed (Participants) | 80 | 81 | 80 | 14 | 14 | 58
  Weight >=5% DFB | 5 | 5 | 7 | 0 | 0 | 4
  Weight >=5% IFB: number analyzed (Participants) | 80 | 81 | 80 | 14 | 14 | 58
  Weight >=5% IFB | 5 | 31 | 27 | 7 | 6 | 15

4. Secondary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Criteria for potentially clinically significant ECG abnormalities:
  * PR Interval: >200 millisecond (ms); >200 ms and IFB >=25%; >220 ms; >220 ms and IFB >=25%; >240 ms; >240 ms and IFB >=25%
  * QRS Interval: >110 ms; >110 ms and IFB >=25%; >120 ms; >120 ms and IFB >=25%
  * QT Interval: >500 ms
  * QTc Bazett (QTc B): >450 ms; 480 ms; 500 ms; IFB >30 and <=60 ms; IFB >60 ms
  * QTc Fridericia (QTc F): >450 ms; 480 ms; 500 ms; IFB >30 and <=60 ms; IFB >60 ms
Time Frame: as for outcome 2
Population: Analysis was performed on safety population.
Measure: Number; unit: participants
Arm/Group | Placebo | Sarilumab 150 mg/150 mg | Sarilumab 200 mg/200 mg | Placebo/Sarilumab 150 mg | Placebo/Sarilumab 200 mg | Sarilumab Rescue
Number analyzed (Participants) | 81 | 81 | 80 | 14 | 15 | 58
participants
  PR Interval >200 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  PR Interval >200 ms | 6 | 9 | 5 | 0 | 2 | 6
  PR Interval >200 ms and IFB >=25%: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  PR Interval >200 ms and IFB >=25% | 0 | 1 | 0 | 0 | 0 | 0
  PR Interval >220 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  PR Interval >220 ms | 3 | 4 | 2 | 0 | 1 | 2
  PR Interval >220 ms and IFB >=25%: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  PR Interval >220 ms and IFB >=25% | 0 | 1 | 0 | 0 | 0 | 0
  PR Interval >240 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  PR Interval >240 ms | 2 | 1 | 0 | 0 | 1 | 2
  PR Interval >240 ms and IFB >=25%: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  PR Interval >240 ms and IFB >=25% | 0 | 0 | 0 | 0 | 0 | 0
  QRS Interval >110 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QRS Interval >110 ms | 2 | 2 | 2 | 1 | 1 | 3
  QRS Interval >110 ms and IFB >=25%: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QRS Interval >110 ms and IFB >=25% | 0 | 0 | 0 | 0 | 0 | 1
  QRS Interval >120 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QRS Interval >120 ms | 2 | 2 | 1 | 1 | 1 | 2
  QRS Interval >120 ms and IFB >=25%: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QRS Interval >120 ms and IFB >=25% | 0 | 0 | 0 | 0 | 0 | 1
  QT Interval >500 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QT Interval >500 ms | 1 | 0 | 1 | 0 | 0 | 3
  QTc B >450 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QTc B >450 ms | 12 | 16 | 22 | 2 | 3 | 18
  QTc B >480 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QTc B >480 ms | 0 | 2 | 2 | 0 | 1 | 2
  QTc B >500 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QTc B >500 ms | 0 | 0 | 0 | 0 | 0 | 0
  QTc B IFB >30 and <=60 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QTc B IFB >30 and <=60 ms | 2 | 2 | 2 | 0 | 1 | 5
  QTc B IFB >60 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QTc B IFB >60 ms | 0 | 0 | 0 | 0 | 0 | 0
  QTc F>450 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QTc F>450 ms | 7 | 11 | 14 | 0 | 2 | 12
  QTc F>480 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QTc F>480 ms | 0 | 0 | 0 | 0 | 1 | 1
  QTc F>500 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QTc F>500 ms | 0 | 0 | 0 | 0 | 0 | 0
  QTc F IFB >30 and <=60 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QTc F IFB >30 and <=60 ms | 4 | 4 | 3 | 0 | 1 | 3
  QTc F IFB >60 ms: number analyzed (Participants) | 77 | 81 | 78 | 14 | 15 | 58
  QTc F IFB >60 ms | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Hematological Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Hemoglobin: <=115 g/L (Male[M]) or <=95 g/L (Female[F]); >=185 g/L (M) or >=165 g/L (F); DFB >=20 g/L
  * Hematocrit: <=0.37 v/v (M) or <=0.32 v/v (F); >=0.55 v/v (M) or >=0.5 v/v (F)
  * Red blood cells (RBC): >=6 Tera/L
  * Platelets: <50 Giga/L; >=50 and <100 Giga/L; >=700 Giga/L
  * White blood cells (WBC): <3.0 Giga/L (Non-Black[NB]) or <2.0 Giga/L (Black[B]); >=16.0 Giga/L
  * Neutrophils: <1.5 Giga/L (NB) or <1.0 Giga/L (B); <1.0 Giga/L
  * Lymphocytes: <0.5 Giga/L; >=0.5 Giga/L and < lower limit of normal (LLN); >4.0 Giga/L
  * Monocytes: >0.7 Giga/L
  * Basophils: >0.1 Giga/L
  * Eosinophils: >0.5 Giga/L or >upper limit of normal (ULN) (if ULN >=0.5 Giga/L)
Time Frame: as for outcome 2
Population: Analysis was performed on safety population.
Measure: Number; unit: participants
Groups:
- Sarilumab Rescue: Participants who received either placebo or sarilumab 150 mg or 200 mg and had inadequate response (defined as less than 20% improvement from baseline on 2 consecutive visits (at least 4 weeks apart) in either TJC or SJC, or with any other clear lack of efficacy based on Investigator's judgment) by Week 16, were rescued with open label sarilumab 200 mg q2w treatment up to Week 52.
Arm/Group | Placebo | Sarilumab 150 mg/150 mg | Sarilumab 200 mg/200 mg | Placebo/Sarilumab 150 mg | Placebo/Sarilumab 200 mg | Sarilumab Rescue
Number analyzed (Participants) | 81 | 81 | 80 | 14 | 15 | 58
participants
  Hemoglobin <=115 g/L (M) or <=95 g/L (F) | 9 | 4 | 5 | 0 | 1 | 5
  Hemoglobin >=185 g/L (M) or >=165 g/L (F) | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin DFB >=20 g/L | 4 | 0 | 3 | 0 | 0 | 1
  Hematocrit <=0.37 v/v (M) or <=0.32 v/v (F) | 17 | 10 | 14 | 0 | 3 | 6
  Hematocrit >=0.55 v/v (M) or >=0.5 v/v (F) | 0 | 0 | 0 | 0 | 0 | 0
  RBC >=6 Tera/L | 0 | 0 | 0 | 0 | 0 | 0
  Platelets <50 Giga/L | 0 | 1 | 0 | 0 | 0 | 0
  Platelets >=50 and <100 Giga/L | 0 | 2 | 4 | 0 | 0 | 1
  Platelets >=700 Giga/L | 1 | 0 | 0 | 0 | 0 | 0
  WBC <3.0 Giga/L (NB) or <2.0 Giga/L (B) | 0 | 30 | 23 | 5 | 6 | 17
  WBC >=16.0 Giga/L | 0 | 5 | 5 | 0 | 0 | 2
  Neutrophils <1.5 Giga/L (NB) or <1.0 Giga/L (B) | 0 | 31 | 24 | 5 | 6 | 18
  Neutrophils <1.0 Giga/L | 0 | 11 | 6 | 3 | 0 | 8
  Lymphocytes <0.5 Giga/L | 3 | 6 | 3 | 1 | 2 | 1
  Lymphocytes >=0.5 Giga/L and <LLN | 23 | 29 | 32 | 4 | 2 | 18
  Lymphocytes >4.0 Giga/L | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes >0.7 Giga/L | 9 | 10 | 7 | 0 | 2 | 3
  Basophils >0.1 Giga/L | 6 | 11 | 9 | 1 | 0 | 9
  Eosinophils>0.5 Giga/L or >ULN(if ULN>=0.5 Giga/L) | 1 | 2 | 1 | 1 | 0 | 2

6. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Metabolic Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Glucose: <=3.9 mmol/L and <LLN; >=11.1 mmol/L unfasted or >=7 mmol/L fasted
  * Hemoglobin A1c (HbA1c): >8%
  * Total cholesterol: >=6.2 mmol/L; >=7.74 mmol/L
  * LDL cholesterol: >=4.1 mmol/L; >=4.9 mmol/L
  * Triglycerides: >=4.6 mmol/L; >=5.6 mmol/L
Time Frame: as for outcome 2
Population: Analysis was performed on safety population.
Measure: Number; unit: participants
Arm/Group | Placebo | Sarilumab 150 mg/150 mg | Sarilumab 200 mg/200 mg | Placebo/Sarilumab 150 mg | Placebo/Sarilumab 200 mg | Sarilumab Rescue
Number analyzed (Participants) | 81 | 81 | 80 | 14 | 15 | 58
participants
  Glucose <=3.9 mmol/L and <LLN | 0 | 0 | 2 | 1 | 1 | 2
  Glucose>=11.1 mmol/L unfasted or >=7 mmol/L fasted | 3 | 8 | 4 | 0 | 0 | 1
  HbA1c >8%: number analyzed (Participants) | 79 | 81 | 78 | 14 | 15 | 58
  HbA1c >8% | 0 | 0 | 0 | 0 | 0 | 0
  Total cholesterol >=6.2 mmol/L | 9 | 40 | 32 | 4 | 2 | 17
  Total cholesterol >=7.74 mmol/L | 0 | 7 | 5 | 0 | 1 | 3
  LDL cholesterol >=4.1 mmol/L | 3 | 20 | 17 | 3 | 1 | 7
  LDL cholesterol >=4.9 mmol/L | 0 | 4 | 6 | 0 | 1 | 2
  Triglycerides >=4.6 mmol/L | 0 | 0 | 3 | 0 | 1 | 2
  Triglycerides >=5.6 mmol/L | 0 | 0 | 3 | 0 | 1 | 2

7. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Electrolytes
Description: Criteria for potentially clinically significant abnormalities:
  * Sodium: <=129 mmol/L; >=160 mmol/L
  * Potassium: <3 mmol/L; >=5.5 mmol/L
  * Chloride: <80 mmol/L; >115 mmol/L
Time Frame: as for outcome 2
Population: Analysis was performed on safety population.
Measure: Number; unit: participants
Arm/Group | Placebo | Sarilumab 150 mg/150 mg | Sarilumab 200 mg/200 mg | Placebo/Sarilumab 150 mg | Placebo/Sarilumab 200 mg | Sarilumab Rescue
Number analyzed (Participants) | 81 | 81 | 80 | 14 | 15 | 58
participants
  Sodium <=129 mmol/L | 0 | 0 | 1 | 0 | 0 | 0
  Sodium >=160 mmol/L | 0 | 0 | 1 | 0 | 0 | 1
  Potassium <3 mmol/L | 0 | 0 | 1 | 0 | 0 | 0
  Potassium >=5.5 mmol/L | 0 | 0 | 2 | 0 | 1 | 0
  Chloride <80 mmol/L | 0 | 0 | 0 | 0 | 0 | 0
  Chloride >115 mmol/L | 0 | 0 | 0 | 0 | 0 | 1

8. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Renal Function Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Creatinine: >=150 micromol/L; >=30% change from baseline; >=100% change from baseline
  * Creatinine clearance: <15 mL/min; >=15 to <30 mL/min; >=30 to < 60 mL/min; >=60 to <90 mL/min
  * Blood urea nitrogen: >=17 mmol/L
  * Uric acid: <120 micromol/L; >408 micromol/L
Time Frame: as for outcome 2
Population: Analysis was performed on safety population.
Measure: Number; unit: participants
Arm/Group | Placebo | Sarilumab 150 mg/150 mg | Sarilumab 200 mg/200 mg | Placebo/Sarilumab 150 mg | Placebo/Sarilumab 200 mg | Sarilumab Rescue
Number analyzed (Participants) | 81 | 81 | 80 | 14 | 15 | 58
participants
  Creatinine >=150 micromol/L | 0 | 1 | 1 | 0 | 1 | 0
  Creatinine >=30% change from baseline | 5 | 18 | 22 | 0 | 4 | 17
  Creatinine >=100% change from baseline | 0 | 1 | 1 | 0 | 1 | 0
  Creatinine clearance <15 mL/min | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine clearance >=15 to <30 mL/min | 0 | 1 | 0 | 0 | 1 | 0
  Creatinine clearance >=30 to <60 mL/min | 6 | 12 | 14 | 0 | 2 | 7
  Creatinine clearance >=60 to <90 mL/min | 41 | 45 | 42 | 7 | 5 | 35
  Blood urea nitrogen >=17 mmol/L | 0 | 0 | 0 | 0 | 1 | 0
  Uric acid <120 micromol/L | 0 | 1 | 2 | 0 | 0 | 0
  Uric acid >408 micromol/L | 8 | 13 | 14 | 3 | 3 | 5

9. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Liver Function Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Alanine Aminotransferase (ALT): >1 ULN and <=1.5 ULN; >1.5 ULN and <=3 ULN; >3 ULN and <=5 ULN; >5 ULN and <=10 ULN; >10 ULN and <=20 ULN; >20 ULN
  * Aspartate aminotransferase (AST): >1 ULN and <=1.5 ULN; >1.5 ULN and <=3 ULN; >3 ULN and <=5 ULN; >5 ULN and <=10 ULN; >10 ULN and <=20 ULN; >20 ULN
  * Alkaline phosphatase: >1.5 ULN
  * Total bilirubin (TBILI): >1.5 ULN; >2 ULN
  * Conjugated bilirubin (CBILI): >1.5 ULN; >2 ULN
  * Unconjugated bilirubin: >1.5 ULN; >2 ULN
  * ALT and TBILI: ALT >3 ULN and TBILI >2 ULN
  * CBILI and TBILI: CBILI >35% TBILI and TBILI >1.5 ULN
  * Albumin: <=25 g/L
Time Frame: For placebo arm: Baseline up to Week 24; For sarilumab 150 mg/150 mg, sarilumab 200 mg/200 mg and sarilumab rescue arm : Baseline up to Week 58; For placebo/sarilumab 150 mg and placebo/sarilumab 200 mg arm: Week 25 up to Week 58
Population: Analysis was performed on safety population.
Measure: Number; unit: participants
Arm/Group | Placebo | Sarilumab 150 mg/150 mg | Sarilumab 200 mg/200 mg | Placebo/Sarilumab 150 mg | Placebo/Sarilumab 200 mg | Sarilumab Rescue
Number analyzed (Participants) | 81 | 81 | 80 | 14 | 15 | 58
participants
  ALT >1 ULN and <=1.5 ULN | 3 | 17 | 24 | 3 | 6 | 16
  ALT >1.5 ULN and <=3 ULN | 7 | 24 | 19 | 4 | 4 | 9
  ALT >3 ULN and <=5 ULN | 6 | 11 | 5 | 2 | 0 | 4
  ALT >5 ULN and <=10 ULN | 0 | 1 | 2 | 0 | 1 | 2
  ALT >10 ULN and <=20 ULN | 0 | 0 | 0 | 0 | 0 | 0
  ALT >20 ULN | 0 | 0 | 0 | 0 | 0 | 0
  AST >1 ULN and <=1.5 ULN | 7 | 34 | 32 | 6 | 8 | 22
  AST >1.5 ULN and <=3 ULN | 11 | 18 | 10 | 3 | 1 | 11
  AST >3 ULN and <=5 ULN | 1 | 5 | 2 | 1 | 1 | 3
  AST >5 ULN and <=10 ULN | 0 | 0 | 1 | 0 | 0 | 0
  AST >10 ULN and <=20 ULN | 0 | 0 | 0 | 0 | 0 | 0
  AST >20 ULN | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase >1.5 ULN | 0 | 2 | 0 | 0 | 0 | 0
  TBILI >1.5 ULN | 0 | 1 | 2 | 1 | 0 | 3
  TBILI >2 ULN | 0 | 0 | 1 | 0 | 0 | 1
  CBILI >1.5 ULN | 0 | 0 | 0 | 0 | 0 | 1
  CBILI >2 ULN | 0 | 0 | 0 | 0 | 0 | 1
  Unconjugated bilirubin >1.5 ULN | 0 | 0 | 1 | 0 | 0 | 1
  Unconjugated bilirubin >2 ULN | 0 | 0 | 0 | 0 | 0 | 0
  ALT >3 ULN and TBILI >2 ULN | 0 | 0 | 0 | 0 | 0 | 0
  CBILI >35% TBILI and TBILI >1.5 | 0 | 0 | 0 | 0 | 0 | 1
  Albumin <=25 g/L | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For placebo arm: Baseline up to Week 24; For sarilumab 150 mg/150 mg, sarilumab 200 mg/200 mg and sarilumab rescue arm: Baseline up to Week 58; For placebo/sarilumab 150 mg and placebo/sarilumab 200 mg arm: Week 25 up to Week 58.
Description: Reported AEs are treatment-emergent AEs that is AEs that developed or worsened or became serious during double-blind on-treatment period, single-blind on-treatment period up to 6-week post-treatment follow-up period (up to Week 58).
Arm/Group | Placebo | Sarilumab 150 mg/150 mg | Sarilumab 200 mg/200 mg | Placebo/Sarilumab 150 mg | Placebo/Sarilumab 200 mg | Sarilumab Rescue
Serious Adverse Events (participants affected / at risk) | 6/81 | 8/81 | 5/80 | 0/14 | 2/15 | 4/58
Other Adverse Events (participants affected / at risk) | 35/81 | 67/81 | 59/80 | 12/14 | 13/15 | 48/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Sarilumab 150 mg/150 mg (N=81) | Sarilumab 200 mg/200 mg (N=80) | Placebo/Sarilumab 150 mg (N=14) | Placebo/Sarilumab 200 mg (N=15) | Sarilumab Rescue (N=58)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infective myositis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Sarilumab 150 mg/150 mg (N=81) | Sarilumab 200 mg/200 mg (N=80) | Placebo/Sarilumab 150 mg (N=14) | Placebo/Sarilumab 200 mg (N=15) | Sarilumab Rescue (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 10 | 9 | 2 | 1 | 6
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Anal erosion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 2 | 2 | 3 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 2 | 4
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1 | 0
Lip erosion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 4 | 0 | 0 | 5
Stomatitis (Gastrointestinal disorders) | 3 | 6 | 8 | 2 | 1 | 7
Injection site erythema (General disorders) | 0 | 8 | 7 | 1 | 0 | 5
Injection site pruritus (General disorders) | 0 | 5 | 4 | 1 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 8 | 7 | 0 | 0 | 4
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 2 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 4 | 1 | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 5 | 1 | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 2 | 6 | 0 | 0 | 3
Gingivitis (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 1 | 2 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 12 | 27 | 23 | 5 | 4 | 19
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 2 | 0 | 2 | 1 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 4 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 4 | 2 | 0 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 8 | 7 | 0 | 0 | 6
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1 | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 7 | 4 | 3 | 0 | 3
Neutrophil count decreased (Investigations) | 0 | 2 | 0 | 1 | 0 | 3
White blood cell count decreased (Investigations) | 0 | 4 | 2 | 0 | 0 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 0 | 1 | 3
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 7 | 4 | 1 | 0 | 3
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 4 | 5 | 0 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.